CLINICAL TRIAL: NCT04544137
Title: Evaluation and Enhancement of the Summer Food Service Program in Youth From an Urban, Low-resource Community
Brief Title: Summer Food Service Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 207716
Record Dates: First submitted 2020-09-03; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Pediatric Obesity; Exercise
Keywords: Summer; Physical Activity; Health disparities
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research staff who completes assessments will not be aware of random assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BOKS + SFSP (Experimental): Children randomized to the BOKS + SFSP will be invited to attend the one-hour BOKS program four days per week for eight weeks during the summer. The BOKS program will be run by Lifespan employed staff in the hour before the SFSP lunch service at two community locations.
  Interventions: Behavioral: BOKS
- SFSP (No Intervention): Children randomized to the SFSP alone group will be asked to participate in the SFSP as they would have otherwise.

INTERVENTIONS:
Behavioral: BOKS — BOKS is an evidence-based physical activity program developed by Reebok to get kids active and establish a lifelong commitment to health and fitness. It was originally developed and tested as a 12-week program offered before or after school. In the present study, BOKS will be offered four days per week for eight weeks over the summer at a public park in one low-income community. The program will run one-hour prior to lunch service by the USDA's Summer Food Service Program. The BOKS curriculum includes lesson plans for 40-45 minute classes that follow the same daily format and focus on a functional fitness skill of the week (squat, plank, push up, etc) and engage participants in team-oriented games.
  Arms: BOKS + SFSP

SUMMARY:
This pilot trial is designed to test the acceptability and preliminary efficacy of offering the BOKS program, an evidence-based physical activity curriculum that engages school-age children in moderate to vigorous physical activity for one hour daily, alongside the USDA's Summer Food Service Program (SFSP) during the summer. Eighty children, ages 6-12 years and from low-income households, will be randomized to participate in the BOKS + SFSP program or to the SFSP alone. We anticipate that the BOKS program will not only provide increased physical activity for the participants, but that it will help to promote participation in the SFSP given that it will be offered in the same location directly before the SFSP lunches are served.

DETAILED DESCRIPTION:
Youth from low-resource communities are disproportionately affected by childhood obesity, independent of race and ethnicity. A time of particular vulnerability for excess weight gain in low-income youth is the summer. Findings from three separate low-income populations show that BMI z-scores (BMIz) decrease during the school year and increase during the summer in this population. To address this and aid in national obesity prevention efforts, the Institute of Medicine and the White House Task Force on Childhood Obesity recommend increased access to the Summer Food Service Program (SFSP), a federally-funded program that provides a free, healthy lunch meal to youth during the summer. However, participation in the SFSP is low. Based on qualitative work with families from low-income communities, this pilot trial is designed to test the acceptability and and preliminary efficacy of the BOKS program, an evidence-based physical activity curriculum that engages school-age children in moderate to vigorous physical activity for one hour daily, when offered alongside the USDA's Summer Food Service Program during the summer. Specifically, 80 children, ages 6-12 years and from low-income households, will be randomized to participate in the BOKS + SFSP program or to the SFSP alone. To test acceptability of the combined program versus the SFSP alone, we will compare SFSP participation (attendance) across groups. Additionally, we will examine physical fitness levels in both groups to determine if participation in the BOKS program prevents the loss of fitness gains achieved during the school year.

ELIGIBILITY:
Inclusion Criteria:

* Reside in the low-income, Rhode Island community where BOKS program is offered
* Quality for free meals as part of the NSLP, which is equivalent to a family of four having an annual income less than $43,568 in the state of Rhode Island.
* Ages 6-12 years
* Ability of the child to speak, read and write English (for purposes of the focus groups and intervention)
* Agreement to randomization

Exclusion Criteria:

* Inability to participate in routine physical activity

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Acceptability of the BOKS + SFSP Programs | 8 weeks
  Attendance in the SFSP

SECONDARY OUTCOMES:
Respiratory Fitness | 8 weeks
  Pacer Test
Excess Summer Weight gain | 8 weeks
  Change in BMIz

CONTACTS AND LOCATIONS:
Locations (1):
- Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No